CLINICAL TRIAL: NCT01411501
Title: Efficacy and Safety of Acupuncture for Functional Constipation: a Multi-center Randomized Controlled Trial
Brief Title: Efficacy and Safety of Acupuncture for Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guangan'men Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011CB505202
Record Dates: First submitted 2011-07-28; First posted 2011-08-08 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Constipation
Keywords: Acupuncture; Functional constipation
MeSH Terms: conditions — Constipation | interventions — Acupuncture Therapy; Moxibustion; mosapride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acupuncture at ST25 and BL25 (Experimental): the points formula of back-shu point combination with front-mu point.
  Interventions: Other: acupuncture
- Acupuncture at LI11 and ST37 (Experimental): the points formula of He-points
  Interventions: Other: acupuncture
- Acupuncture at ST25, BL25, LI11 and ST37 (Experimental): the formula of He-point,back-shu point and front-mu point
  Interventions: Other: acupuncture
- medicine (Active Comparator): oral use of mosapride citrate
  Interventions: Drug: mosapride citrate

INTERVENTIONS:
Other: acupuncture — Thrust and lift the needle to achieve De Qi. After being needled, the points will be punctured again using auxiliary needles 2 mm lateral to the first needle, and to a depth of 2 mm without manual stimulation. Put the electric stimulator on the pair of needles with a continuous wave, 20Hz. The current intensity is increased to the patients' maximum tolerance and then slightly reduced to a bearable level (0.1-1.0 mA).
  Huatuo Brand needle (φ0.30×25mm,φ0.30×40mm,φ0.30×50mm, produced by Suzhou Medical Appliance Factory) and G6805-1A electro-acupuncture apparatus(produced by Shanghai Huayi Medical Instrument Co. Ltd.) will be used.
  Five sessions/week in the first 2 weeks, three sessions/week for in the last 2 weeks.
  Other Names: acupuncture and moxibustion
  Arms: Acupuncture at LI11 and ST37; Acupuncture at ST25 and BL25; Acupuncture at ST25, BL25, LI11 and ST37
Drug: mosapride citrate — 4-week oral use of mosapride citrate, 5mg, three times daily 0.5 hour before meal
  Other Names: mosapride citrate,made in China
  Arms: medicine

SUMMARY:
A multi-center clinical trial done recently by us(NCT00508482) shows that needling on ST25 has the same effect as lactulose in unaided self-defecation frequency of a week and has better effect in symptoms improvement (in press). The object is to evaluate whether acupuncture is effective for functional constipation. As an explanatory research, it took one single point as its intervention and sham acupuncture as its control group (patients were blinded). On the basis of its confirmed effect, we are taking a pragmatic randomized controlled trial to further evaluate whether acupuncture is more effective than routine treatment. Acupuncture prescriptions used in this trial are individually prescribed according to syndrome differentiation, which can improve clinical effect. .

DETAILED DESCRIPTION:
functional constipation,acupuncture,effects and safety,pragmatic RCT

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been diagnosed with functional constipation according to Rome Ⅲ criteria
* Patients who are aged 18-75 years old
* Stop medication or acupuncture (if any) 1 week before randomization and uninvolved in other trials
* Sign the informed consent out of one's own will

Exclusion Criteria:

* Secondary constipation
* Patients with consciousness impairment, psychotic patients or patients unable to express clearly
* Patients with malignant tumor in progressive stage, severe wasting disease and liable to be infected and bleed
* Patients with severe cardiovascular disease, hepatic injury, renal damage, digestive disease or hematological diseases
* Women in pregnancy and lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LIU Zhishun, phD, Study Chair — Guang'an Men Hospital Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- No.5 Beixiange Street, Xuanwu District, Beijing, China

REFERENCES:
- [Derived] Li Y, Zheng H, Zeng F, Zhou SY, Zhong F, Zheng HB, Chen M, Jing XH, Cai YY, Jia BH, Zhu B, Liu ZS. Use acupuncture to treat functional constipation: study protocol for a randomized controlled trial. Trials. 2012 Jul 3;13:104. doi: 10.1186/1745-6215-13-104. PMID 22759406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited through the inpatients and outpatients settings in the 8 hospitals.We also recruited the participants through television and newspapers advertisements.
Pre-assignment Details: Nine enrolled participants refused to join in the trial after signing the informed consent. So they were excluded from the trial.
Groups:
- Acupuncture at ST25 and BL25: the points formula of back-shu point combination with front-mu point.
  acupuncture: Thrust and lift the needle to achieve De Qi. After being needled, the points will be punctured again using auxiliary needles 2 mm lateral to the first needle, and to a depth of 2 mm without manual stimulation. Put the electric stimulator on the pair of needles with a continuous wave, 20Hz. The current intensity is increased to the patients' maximum tolerance and then slightly reduced to a bearable level (0.1-1.0 mA).
  Huatuo Brand needle (φ0.30×25mm,φ0.30×40mm,φ0.30×50mm, produced by Suzhou Medical Appliance Factory) and G6805-1A electro-acupuncture apparatus(produced by Shanghai Huayi Medical Instrument Co. Ltd.) will be used.
  Five sessions/week in the first 2 weeks, three sessions/week for in the last 2 weeks.
- Acupuncture at LI11 and ST37: the points formula of He-points
  acupuncture: Thrust and lift the needle to achieve De Qi. After being needled, the points will be punctured again using auxiliary needles 2 mm lateral to the first needle, and to a depth of 2 mm without manual stimulation. Put the electric stimulator on the pair of needles with a continuous wave, 20Hz. The current intensity is increased to the patients' maximum tolerance and then slightly reduced to a bearable level (0.1-1.0 mA).
  Huatuo Brand needle (φ0.30×25mm,φ0.30×40mm,φ0.30×50mm, produced by Suzhou Medical Appliance Factory) and G6805-1A electro-acupuncture apparatus(produced by Shanghai Huayi Medical Instrument Co. Ltd.) will be used.
  Five sessions/week in the first 2 weeks, three sessions/week for in the last 2 weeks.
- Acupuncture at ST25, BL25, LI11 and ST37: the formula of He-point,back-shu point and front-mu point
  acupuncture: Thrust and lift the needle to achieve De Qi. After being needled, the points will be punctured again using auxiliary needles 2 mm lateral to the first needle, and to a depth of 2 mm without manual stimulation. Put the electric stimulator on the pair of needles with a continuous wave, 20Hz. The current intensity is increased to the patients' maximum tolerance and then slightly reduced to a bearable level (0.1-1.0 mA).
  Huatuo Brand needle (φ0.30×25mm,φ0.30×40mm,φ0.30×50mm, produced by Suzhou Medical Appliance Factory) and G6805-1A electro-acupuncture apparatus(produced by Shanghai Huayi Medical Instrument Co. Ltd.) will be used.
  Five sessions/week in the first 2 weeks, three sessions/week for in the last 2 weeks.
Period: Overall Study
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Started | 168 | 172 | 165 | 170
Completed | 158 | 166 | 159 | 163
Not Completed | 10 | 6 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine | Total
Number analyzed (Participants) | 168 | 172 | 165 | 170 | 675
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (17.4) | 39.9 (16.8) | 40.7 (16.8) | 40.6 (16.7) | 40.1 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 140 | 138 | 142 | 548
  Male | 40 | 32 | 27 | 28 | 127
Region of Enrollment [Number; unit: participants]
  China | 168 | 172 | 165 | 170 | 675
Duration of functional constipation [Mean (Standard Deviation); unit: months] | 7.0 (6.8) | 6.3 (6.5) | 5.6 (4.3) | 5.8 (4.6) | 6.2 (5.56)
Received Traditional Chinese Medicine therapies [Number; unit: participants]
  Acupuncture | 7 | 9 | 7 | 3 | 26
  Herbs | 38 | 48 | 43 | 44 | 173
  Both | 7 | 5 | 8 | 5 | 25
  Neither | 116 | 110 | 107 | 118 | 451
SBMs [Mean (Standard Deviation); unit: times per week] — SBMs, spontaneous bowel movements.
  times per week | 2.7 (1.9) | 2.5 (1.7) | 2.9 (2.0) | 2.9 (2.8) | 2.8 (2.1)
Bristol scale [Mean (Standard Deviation); unit: units on a scale] — Bristol stool scale provides illustration of seven stool types. It ranges from 1 to 7 with the meaning that 1 referring to separate hard lumps and 7 referring to watery, no solid pieces. For patients with constipation, a higher score means a better outcome.
  units on a scale | 2.8 (1.3) | 2.9 (1.4) | 3.0 (1.5) | 2.7 (1.4) | 2.9 (1.8)
Degree of straining during defecation [Number; unit: participants] — This outcome describes how much effort the patients with while defecating. It ranges from 0 to 3. Zero means defecating with no effort and 3 means defecating with great effort. A 0 score is considered a better than 3 for outcome. Patients score for themselves according to their own feelings.
  participants
    0 | 5 | 8 | 9 | 5 | 27
    1 | 63 | 60 | 68 | 59 | 250
    2 | 68 | 69 | 58 | 72 | 267
    3 | 30 | 35 | 28 | 31 | 124
    no defecation | 2 | 0 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change of the SBMs From Baseline at Week 4
Description: [average number of spontaneous bowel movements in a week at week 4]-[average number of spontaneous bowel movements in a week at baseline]
Time Frame: baseline and at 4 weeks
Measure: Mean (95% Confidence Interval); unit: times per week
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Number analyzed (Participants) | 168 | 172 | 165 | 170
times per week | 2.7 [2.3 to 3.0] | 2.7 [2.3 to 3.1] | 2.2 [1.9 to 2.5] | 2.4 [2.0 to 2.9]
Statistical Analysis 1: Comparison: Acupuncture at ST25 and BL25 vs Acupuncture at LI11 and ST37 vs Acupuncture at ST25, BL25, LI11 and ST37 vs Medicine; Test type: Superiority or Other; p = 0.352, ANCOVA

2. Secondary Outcome: Change From Baseline in the Bristol Stool Scale at the 4th Week
Description: Bristol stool scale provides illustration of seven stool types. It ranges from 1 to 7 with the meaning that 1 referring to separate hard lumps and 7 referring to watery, no solid pieces. For patients with constipation, a higher score means a better outcome. This outcome means the Bristol Stool Scale at the 4th week-the Bristol Stool Scale at baseline.
Time Frame: baseline and at 4 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Number analyzed (Participants) | 168 | 172 | 165 | 170
units on a scale | 3.9 [3.7 to 4.1] | 3.9 [3.8 to 4.1] | 3.9 [3.7 to 4.1] | 3.9 [3.7 to 4.1]
Statistical Analysis 1: Comparison: Acupuncture at ST25 and BL25 vs Acupuncture at LI11 and ST37 vs Acupuncture at ST25, BL25, LI11 and ST37 vs Medicine; Test type: Superiority or Other; p = 0.968, ANCOVA

3. Secondary Outcome: Change From Baseline in Difficulty Degree of Defecation at the 4th Week
Description: This outcome describes how much effort the patients with while defecating.It ranges from 0 to 3.
  0-Without difficulty
  1. Defecation straining
  2. Severe defecation straining
  3. Defecation with the help of hands, A 0 is considered better than 3 for outcome. Patients score for themselves according to their own feelings.
  [the average score of one week at the 4th week]-[the average score of one week at baseline]
Time Frame: baseline and at 4 weeks
Measure: Number; unit: participants
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Number analyzed (Participants) | 158 | 167 | 161 | 164
participants
  0 | 40 | 41 | 33 | 36
  1 | 69 | 78 | 76 | 76
  2 | 33 | 36 | 38 | 43
  3 | 16 | 12 | 14 | 9
Statistical Analysis 1: Comparison: Acupuncture at ST25 and BL25 vs Acupuncture at LI11 and ST37 vs Acupuncture at ST25, BL25, LI11 and ST37 vs Medicine; Test type: Superiority or Other; p = 0.841, Kruskal-Wallis

4. Secondary Outcome: Changes of the SBMs From Baseline at Week 8
Description: [average number of spontaneous bowel movements in a week at week 8]-[average number of spontaneous bowel movements in a week at baseline]
Time Frame: baseline and at 8 weeks
Measure: Mean (95% Confidence Interval); unit: times per week
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Number analyzed (Participants) | 168 | 172 | 165 | 170
times per week | 2.3 [1.9 to 2.7] | 2.4 [2.1 to 2.7] | 2.1 [1.7 to 2.5] | 1.4 [1.0 to 1.8]
Statistical Analysis 1: Comparison: Acupuncture at ST25 and BL25 vs Acupuncture at LI11 and ST37 vs Acupuncture at ST25, BL25, LI11 and ST37 vs Medicine; Test type: Superiority or Other; p = 0.005, ANCOVA

5. Secondary Outcome: Change From Baseline in the Bristol Stool Scale at the 8th Week
Description: Bristol stool scale provides illustration of seven stool types. It ranges from 1 to 7 with the meaning that 1 referring to separate hard lumps and 7 referring to watery, no solid pieces. For patients with constipation, a higher score means a better outcome. This outcome means the Bristol Stool Scale at the 8th week-the Bristol Stool Scale at baseline.
Time Frame: baseline and at 8 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Number analyzed (Participants) | 168 | 172 | 165 | 170
units on a scale | 3.4 [3.2 to 3.6] | 3.6 [3.5 to 3.8] | 3.4 [3.2 to 3.6] | 3.1 [2.9 to 3.3]
Statistical Analysis 1: Comparison: Acupuncture at ST25 and BL25 vs Acupuncture at LI11 and ST37 vs Acupuncture at ST25, BL25, LI11 and ST37 vs Medicine; Test type: Superiority or Other; p = 0.198, ANCOVA

6. Secondary Outcome: Change From Baseline in Difficulty Degree of Defecation at the 8th Week
Description: This outcome describes how much effort the patients with while defecating. It ranges from 0 to 3.
  0-Without difficulty
  1. Defecation straining
  2. Severe defecation straining
  3. Defecation with the help of hands, A 0 is considered better than 3 for outcome. Patients score for themselves according to their own feelings.
  [the average score of one week at the 8th week]-[the average score of one week at baseline]
Time Frame: baseline and at 8 weeks
Measure: Number; unit: participants
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Number analyzed (Participants) | 158 | 166 | 159 | 163
participants
  0 | 45 | 46 | 40 | 36
  1 | 75 | 88 | 83 | 67
  2 | 29 | 25 | 28 | 44
  3 | 9 | 7 | 8 | 16
Statistical Analysis 1: Comparison: Acupuncture at ST25 and BL25 vs Acupuncture at LI11 and ST37 vs Acupuncture at ST25, BL25, LI11 and ST37 vs Medicine; Test type: Superiority or Other; p = 0.035, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Acupuncture at ST25 and BL25 | Acupuncture at LI11 and ST37 | Acupuncture at ST25, BL25, LI11 and ST37 | Medicine
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/172 | 0/165 | 0/170
Other Adverse Events (participants affected / at risk) | 3/168 | 3/172 | 6/165 | 6/170
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture at ST25 and BL25 (N=168) | Acupuncture at LI11 and ST37 (N=172) | Acupuncture at ST25, BL25, LI11 and ST37 (N=165) | Medicine (N=170)
Eye discomfort (Eye disorders) | 0 | 1 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Common cold (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3
Joint pains (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 0
Fundus hemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Unblinding of participants in the acupuncture and mosapride groups;an insufficient duration to assess the long term effect or risks;a missing assessment of electrocardiograms for possible cardiovascular harm of mosapride

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No